CLINICAL TRIAL: NCT05605756
Title: BOTOX Effects on Seizure Severity and Susceptibility
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Failure to recruit subjects.
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Rami Burstein, John Hedley-Whyte Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P000215
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Drug-resistant Focal Seizure
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Botox therapy effects on seizure (Experimental)
  Interventions: Drug: OnabotulinumtoxinA 145 UNT [Botox]

INTERVENTIONS:
Drug: OnabotulinumtoxinA 145 UNT [Botox] — Botulinum A toxin injection: Will follow the FDA-approved guideline of the treatment of chronic migraine. The following modifications are planned: (a) Total units 145 instead of 155. (b) Number of injection sites 29 instead of 31. (c) the 6 injection sites in the trapezius muscle will be eliminated as they are irrelevant to our attempt to reduce seizure events. Instead, 4 injections will be made subcutaneously along the superior sagittal suture (see figures below), where no muscles exist and thus no muscle weakness is likely. This dose (145 Units) is well below the FDA-approved guideline on safety for adolescents and adults (no more than 10 Units/Kg or a total of 340 Units).
  Botox injections will take place in the BIDMC Headache Clinic which is a part of the Arnold Pain center at 1 Brookline Place. Injections will be administered by Dr. Sait Ashina, the Director of the Headache Clinic.
  Other Names: BOTOX

SUMMARY:
The purpose of this research is to determine whether BOTOX injections will reduce seizure frequency and severity. We chose to test its effects on epilepsy because epilepsy and migraine have common features so, are often treated with common drugs.

DETAILED DESCRIPTION:
Goals:

The purpose of this study is to determine whether BOTOX injections into the scalp raise seizure threshold such that focal seizures are less likely to occur, and less likely to generalize.

Objectives:

1. To test whether scalp BOTOX injections mitigate seizure frequency or seizure severity. This objective will be tested using a prospective clinical observation in patients with focal epilepsy (see definitions below)
2. To test whether quantitative measures of seizures susceptibility (cortical excitability) are altered by scalp BOTOX injections. This objective will be tested using 24-hour ambulatory scalp EEG recording and transcranial magnetic stimulation (TMS) with simultaneous EEG/EMG a noninvasive tool to measure cortical excitability (Tsuboyama et al 2019).

Clarification of terminology:

* Focal seizures are seizures that arise in one area of the brain.
* Focal seizures with impaired awareness are seizures that arise in one area of the brain, and often spread to areas associated with conscious experience (i.e., are associated with alteration of awareness).
* Focal to bilateral tonic clonic seizures are seizures that arise in one brain region and spread to the entire forebrain, bilaterally and manifest as a convulsion.
* Primary generalized seizures are seizure that arise simultaneously in both hemispheres.

Overall Study Design:

In a single-center open-label study, patients with pharmaco-resistant focal epilepsy will undergo 8-week seizure monitoring and baseline 24-hour ambulatory EEG and TMS-EEG-EMG. This period will take place between day 1 and day 59 (see flowchart). Each patient will then be injected with BOTOX (145 units) according to the FDA-approved paradigm for the treatment of migraine, plus injections along the sagittal suture. Seizure diary will be maintained for the duration of the study. EEG and TMS-EEG-EMG will be repeated 21 days, when BOTOX effects usually begin, and 8 weeks after injection, when BOTOX effect are usually at their peak. Data will then be analyzed to measure BOTOX antiepileptic capacity.

Screening and Enrollment Period (1 in-person visit):

Participants will initially be screened in person and written consent will be obtained. Screening will include a review of medical, surgical and seizure history and current medication review. They will be provided instruction on maintaining a daily seizure diary for 8 weeks in order to capture their baseline seizure frequency. If frequency is less than an average of 3 seizures/month or if there is a change in their seizure medication, the participant will be excluded at that time. Due to variability in seizure frequency, the baseline seizure monitoring period may be extended up to an additional 4 weeks.

Baseline and Follow-up EEG and TMS with EEG Assessments (2 visits at each time point - 6 total visits):

Once the participant is fully screened, they will come to BIDMC to be set up with a 24 hour ambulatory EEG. A second study visit will include the TMS with EEG testing (details provided below in "Procedures"). If a participant screens out of being TMS eligible, the participant will still be included and this visit will not occur. These assessments will be repeated 21 and 56 days (+/- 5 days) after the Botox injection. Neuro QOL questionnaires will be completed at baseline, 56 weeks after Botox and the final visit.

PROCEDURES:

-Botulinum A toxin injection: Will follow the FDA-approved guideline of the treatment of chronic migraine. The following modifications are planned: (a) Total units 145 instead of 155. (b) Number of injection sites 29 instead of 31. (c) the 6 injection sites in the trapezius muscle will be eliminated as they are irrelevant to our attempt to reduce seizure events. Instead, 4 injections will be made subcutaneously along the superior sagittal suture (see figures below), where no muscles exist and thus no muscle weakness is likely. This dose (145 Units) is well below the FDA-approved guideline on safety for adolescents and adults (no more than 10 Units/Kg or a total of 340 Units).

Botox injections will take place in the BIDMC Headache Clinic which is a part of the Arnold Pain center at 1 Brookline Place. Injections will be administered by Dr. Sait Ashina, the Director of the Headache Clinic.

EEG: 24-hour ambulatory EEG with 10-20 international system of electrode placement will be obtained at three time points: (1) 1-4 weeks prior to BOTOX injections, (2) 21 days/3 weeks (+/- 5 days) after BOTOX injections, (3) 56 days/8-weeks (+/- 5 days) after BOTOX injection.

TMS: TMS-derived metrics will be obtained at the same three time points as EEG: (1) 1-4 weeks prior to BOTOX injections, (2) 21 days/3 weeks (+/- 5 days) after BOTOX injections, (3) 56 days/8-weeks (+/- 5 days) after BOTOX injection. TMS is a safe, non-invasive method of focal cortical stimulation used to measure the cortical excitation/inhibition (E:I) ratio. A magnetic field is generated by a powerful extracranial magnet that induces intracranial electrical currents over the focal region of stimulation. When coupled with surface EMG electrodes (TMS-EMG), output resultant from stimulation over the motor cortex can be measured as a motor evoked potential (MEP) from a target muscle (most often the abductor pollicis brevis, APB).

All TMS-EMG-EEG sessions will be identical. Subjects will be set up in a chair with an EEG cap and with EMG electrodes placed on both hands for collection of MEPs during stimulation over the bilateral motor cortices (M1). The EEG cap and electromyography (EMG) electrodes will remain in place throughout the TMS session. The session will include resting-state EEG measurements; determination of motor threshold and input-output curve, cortical silent period, single pulse and paired pulse TMS-EEG in up to 8 brain regions (left and right frontal lobes, left and right motor cortex, left and right parietal lobes, and left and right occipital lobes). Each subject will undergo sham stimulation to control for nonspecific effects, such as the auditory evoked potential. The total time of the session will be approximately 4-5 hours.

Seizure Tracking:

All subjects and families will utilize a digital seizure diary (seizuretracker.com), but with the option to use paper diaries instead if they prefer. Proficiency in seizure diary maintenance will be confirmed by study staff during the screening period. Study staff may call the participant to remind them to complete their diary entries and/or to re-educate the participant regarding maintaining the diary. Seizure documentation (frequency, severity, gross description) will be maintained for 8 weeks before and 12 weeks after BOTOX injections.

If participants choose to use the digitial seizure diary, they will be asked to share their information with the study team via the Valet system, by printing reports from SeizureTracker or by visually and verbally (via phone call check-ins) sharing the information that they have documented in their diary, just as they would if they choose to keep a paper diary. It is not possible to download data from the Valet system - the study team will write down and/or direct enter into REDCap the details that the participant shares regarding their diary. Of note, is that SeizureTracker is a very common App that patients with epilepsy routinely use and are familiar with. Participants who choose to join seizuretracker to maintain their diary for the study will be advised to not utilize the Alexa feature and will be instructed to carefully review the features that they can opt out of along with the Terms and Conditions for users. There are participants who may already use seizuretracker prior to engaging in the study, therefore, they will already have made their personal choices regarding use of the program. Lastly, participants will ahv the option of continuing or closing their account at the end of the study.

Study staff will check the seizure diary weekly to make note of frequency as compared to baseline. If a participant has an increase in seizure frequency at or above 100% from baseline over 4 weeks, the study MD will review the seizure tracking and diary, talk with the participant and, per the clinician judgement, may refer the participant to their provider for follow-up. The 4 week time frame is to account for a patient population that has frequent seizures and can experience clusters of seizures and/or can have stressful conditions/triggers that may temporarily increase seizure frequency. In addition, the study team (including the study MD/epileptologist) will review the seizure frequency/diary of all post-Botox injection participants on a weekly basis to identify if a participant is trending in this direction so that the study MD can make a judgement if there is a clinical concern/need to further review the participant's status at any point.

Neuro-QOL:

Participants will be asked to complete components of the standardized Neuro Quality of Life assessment, a self- report tool used to measure health related quality of life in a wide range of neurologic disorders. Participants are asked to score their responses to prompts on a scale of 1-5. The following components will be used in this study (copies of the scales are attached): Ability to Participate in Social Roles, Anxiety , Depression, Emotional and Behavioral Dyscontrol, Fatigue, Positive Affect and Well-Being, Stigma, Satisfaction with Social Roles and Activities, and Cognitive Function.

ELIGIBILITY:
Patients with focal drug-resistant epilepsy (see inclusion and exclusion criteria).

Potential study subjects will be provided an informed consent form (ICF) to review. Those who are interested in participating will provide informed consent and then be screened for eligibility (inclusion/exclusion criteria). Individuals screened as potential study subjects must meet all the following inclusion criteria and none of the following exclusion criteria.

Inclusion criteria:

* Age: 18-85 years, inclusive
* Sex: Males and females
* Pharmaco-resistant focal epilepsy with >3 seizures a month

Exclusion criteria:

* Cranial or scalp surgery within 3 months of recruitment
* Change in antiepileptic medication <2 months before recruitment
* History of status epilepticus within 12 months of recruitment
* History of psychogenic nonepileptic seizures
* History of poor medication compliance
* Any unstable medical condition
* Any psychiatric disorder that could interfere with trial participation
* Substance use disorders within the past six months
* Pregnancy, breastfeeding, or planning a pregnancy during the trial; unable or unwilling to use a reliable form of contraception during the trial - All individuals of childbearing potential will undergo urine pregnancy testing
* TMS exclusion only (If a participant does not meet TMS criteria, they will not be excluded from the study/the TMS assessments will not be completed):

  * Intracranial metal implants (excluding dental fillings) or devices such as pacemaker, medication pump, nerve stimulator, TENS unit, ventriculo-peritoneal shunt unless cleared by the responsible covering TMS MD.
  * Any intracranial lesions or prior brain surgeries other than minor procedures as reviewed and approved by the TMS MD (e.g. history of brain biopsy, depth electrodes, ICP monitoring, intraventricular and subdural drains…)

Exclusion criteria for Botox

* History of botulinum A toxin injection within 3 months of recruitment
* Allergy to botulinum toxin
* Any medical condition that might put participants at increased risk if exposed to onabotulinumtoxinA (e.g. neuromuscular diseases such as myasthenia gravis, Eaton-Lambert Syndrome, amyotrophic lateral sclerosis)
* Use of any headache prophylactic medication within 28 days before start of baseline
* History of "complicated" migraine
* Fibromyalgia
* Use of opioids as acute pain medication
* Skin problems, infections, profound atrophy, or excessive weakness in the target areas of the injection sites
* Concurrent chronic use or chronic use in the 3 months prior to the screening period of muscle relaxants

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
• Reduction in incidence of generalized seizures | 150 days
  Frequency of generalized seizure will be averaged per time blocks as follows: (1) baseline, 8 weeks before botulinum A toxin injection, (2) 0-4 weeks after BOTOX injections, and (3) 5-12 weeks after BOTOX injection
• Reduction in incidence of focal seizures with impaired awareness | 150 days
  Frequency of focal seizures with impaired awareness will be averaged per time blocks as follows: (1) baseline, 8 weeks before botulinum A toxin injection, (2) 0-4 weeks after BOTOX injections, and (3) 5-12 weeks after BOTOX injection

SECONDARY OUTCOMES:
• Reduction in overall seizure frequency | 150days
  Frequency of overall seizure frequency will be averaged per time blocks as follows: (1) baseline, 8 weeks before botulinum A toxin injection, (2) 0-4 weeks after BOTOX injections, and (3) 5-12 weeks after BOTOX injection
• Reduction in net cortical excitability metrics | 150 days
  TMS metrics of rMT, CSP, LICI, and TMS-EEG excitability metrics will each be averaged over at least 20 trials per subject per time block (at baseline, and 3 weeks and 8 weeks after BOTOX injections). Per metric mean values will then be compared by one-way repeated measures ANOVA.
• Improvement in quality-of-life metrics | 150 days
  Blended Neuro-QOL scores will be averaged at baseline, and at the 8-12 week after BOTOX injection period, and compared by paired t-test

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No